CLINICAL TRIAL: NCT05373303
Title: The Clinical Study for Evaluating The Safety And Efficacy Of Epodion® During Maintenance Period Until Evaluation Period On CKD (Chronic Kidney Disease) Patients: An Open Label, Randomized, Active Drug-Comparative, Parallel-Designed, Multi-Center Clinical Study
Brief Title: The Clinical Study for Evaluating The Safety And Efficacy Of Epodion®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PT. Daewoong Infion (Industry)
Collaborators: Equilab International (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DW_EPO401
Record Dates: First submitted 2022-04-26; First posted 2022-05-13 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: open-label, randomized, active drug-comparative, parallel-designed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Drug (Experimental): Recombinant Human Erythropoietin Alfa, dosage : 50 IU/Kg body weight three times per week, and continued to titrated dose closely to achieve baseline Hb level 10-12g/dL
  Interventions: Biological: Recombinant Human Erythropoietin Alpha
- Reference Drug (Active Comparator): Recombinant Human Erythropoietin Alfa, dosage : 50 IU/Kg body weight three times per week, and continued to titrated dose closely to achieve baseline Hb level 10-12g/dL
  Interventions: Biological: Recombinant Human Erythropoietin Alpha

INTERVENTIONS:
Biological: Recombinant Human Erythropoietin Alpha — This study consisted of a screening period (4 weeks), titration period (4~8 weeks) baseline evaluation period (4 weeks), maintenance period (24 weeks), and 4 weeks for the evaluation period. Patients who were eligible in the screening period underwent the titration period. The reference product at an individualized dose 3 times a week through intravenous injection was given and the hemoglobin (Hb) level of the subject was controlled to reach the target range of 10-12 g/dL in the titration period. In the maintenance period, the subjects were randomized and administered with reference product or test product that was done with the same doses regimen during the titration period through intravenous injection
  Arms: Test Drug
Biological: Recombinant Human Erythropoietin Alpha — This study consisted of a screening period (4 weeks), titration period (4~8 weeks) baseline evaluation period (4 weeks), maintenance period (24 weeks), and 4 weeks for the evaluation period. Patients who were eligible in the screening period underwent the titration period. The reference product at an individualized dose 3 times a week through intravenous injection was given and the hemoglobin (Hb) level of the subject was controlled to reach the target range of 10-12 g/dL in the titration period. In the maintenance period, the subjects were randomized and administered with reference product or test product that was done with the same doses regimen during the titration period through intravenous injection
  Arms: Reference Drug

SUMMARY:
The study was conducted to evaluate whether the efficacy and safety profile of recombinant human erythropoietin (rhEPO) manufactured by Daewoong Pharmaceutical Co., Ltd was similar to biological products approved by the drug safety regulatory authority.

DETAILED DESCRIPTION:
This was an open-label, randomized, active drug-comparative, parallel-designed, multi-center study in hemodialysis patients with anemia.

This study consisted of a screening period (4 weeks), titration period (4~8 weeks) baseline evaluation period (4 weeks), maintenance period (24 weeks), and 4 weeks for the evaluation period. Patients who were eligible in the screening period underwent the titration period. The reference product at an individualized dose 3 times a week through intravenous injection was given and the hemoglobin (Hb) level of the subject was controlled to reach the target range of 10-12 g/dL in the titration period. In the maintenance period, the subjects were randomized and administered with reference product or test product that was done with the same doses regimen during the titration period through intravenous injection. The primary endpoints of efficacy evaluation were to demonstrate that treatment of test product was equivalence with the reference product by evaluating Hb level change between baseline (Week 5-8/9-12) and evaluation period (Week 33-36/37-40), while the secondary endpoints were to obtain data mean change in weekly dosage per kg body weight between the baseline period and the evaluation period, to calculate instability rate of Hb level during maintenance and evaluation period as defined when Hb level dropped below 8 g/dL or increased by more than 13 g/dL and to evaluate the Hb and hematocrit (Ht) level during maintenance and evaluation period. The safety evaluation was conducted based on the incidence of the adverse events of both local and systemic reactions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who are at least 18 years old and younger than 75 years of age at the time of screening visit.
* Patients with End-Stage Renal Failure (ESRD) who are chronically receiving hemodialysis and have anemia.
* Patients with a mean baseline Hb concentration within Hb level ≥ 9 g/dL during the screening period.
* Haemodialysis patients with anemia associated with Chronic Kidney Disease (CKD) currently receiving stable maintenance therapy with Epoetin alfa at least once per week
* Adequate iron substitution status (serum ferritin ≥ 100 μg /dl or saturated transferrin levels ≥ 20%).
* Patients who understand the information provided to them or their representatives and may provide written consent.

Exclusion Criteria:

* Contraindication with Epoetin therapy.
* Documented active bleeding in the last 12 weeks prior to screening period.
* Any blood transfusion within the last 2 weeks prior Screening period.
* History of malignancy of any organ system within the last 5 years.
* Patients with uncontrolled hypertension (in case the mean value of diastolic blood pressure as measured 4 times during the baseline observation period is 110 mmHg or more).
* Patients hyporesponsive epoetin treatment or had medical history of experiencing pure red blood cell forming failure after being administered with Epoetin products.
* Known bone marrow fibrosis (osteitis fibrosa cystica).
* Patient with serious cardiovascular disorders: myocardial infarction, patients with congestive heart failure (NYHA class Ⅲ or higher), ischemic vascular disease
* Patient received percutaneous coronary intervention (PCI), or coronary artery bypass grafting (CABG) during the last 6 months prior to screening.
* Patient with the following liver disorder: Patient diagnosed with liver cirrhosis, hepatitis B, or on active treatment hepatitis C, and patients with ALT or AST exceeding the upper limits of the normal level by more than double.
* Patients whose kidney transplant is expected or already planned for survival.
* Secondary anemia to other causes different to the CKD (aplastic anemia, hemolytic anemia, sickle cell anemia, multiple myeloma, leukemia, myelodysplastic syndrome).
* Patients with the following diseases and who are considered unfit to enroll in the clinical study: mental system disease, mental disease, drug intoxication, epilepsy, lung infarction, cerebral infarction, positive HIV antibody, systemic lupus erythematosus, immunosuppressive condition and general infection
* Pregnancy or lactation period in female patients, or women of childbearing potential without an effective method of birth control.
* Patients who were considered unfit for study by the principal investigators or by the co-investigator.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Hb level change | baseline (Week 5-8/9-12) and evaluation period (Week 33-36/37-40).
  Hb level change between Test and Reference Drug

SECONDARY OUTCOMES:
mean change in weekly dosage per kg body weight | baseline (Week 5-8/9-12) and evaluation period (Week 33-36/37-40).
  Dosage for Mean change in mg/Kg Body Weight

OTHER OUTCOMES:
instability rate of Hb (hemoglobin) | maintenance (week 10-14/32-36) and evaluation period (Week 33-36/37-40)
  instability rate of Hb in Percent (%)
Hb (hemoglobin) and hematocrit level | maintenance (week 10-14/32-36) and evaluation period (Week 33-36/37-40)
  Hb (hemoglobin) in gram/desiLiter and hematocrit level in Percent (%)
incidence of adverse event | during the study evaluation from baseline (Week 5-8/9-12) to evaluation period (Week 33-36/37-40)
  incidence of adverse event between Test and Reference Drug

CONTACTS AND LOCATIONS:
Overall Officials: Jonny Jonny, MD, Principal Investigator — Gatot Soebroto Army Hospital, Jakarta
Locations (1):
- Gatot Soebroto Army Hospital, Jakarta, Indonesia

DOCUMENTS (3):
  • Study Protocol (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT05373303/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT05373303/SAP_001.pdf
  • Informed Consent Form (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/03/NCT05373303/ICF_002.pdf